CLINICAL TRIAL: NCT02190279
Title: A Pilot Study of 18F-DCFBC PET/CT in Prostate Cancer
Brief Title: 18F-DCFBC PET/CT in Prostate Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Maria Liza Lindenberg, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 140140; 14-C-0140
Record Dates: First submitted 2014-07-12; First posted 2014-07-15 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Prostatic Neoplasms; Prostate Cancer
Keywords: Prostate Specific Membrane Antigen; Radiolabeled PET Agent; Imaging; NaF
MeSH Terms: conditions — Prostatic Neoplasms | interventions — N-(N-((S)-1,3-Dicarboxypropyl)carbamoyl)-4-(18F)fluorobenzyl-L-cysteine; Sodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Suspected Localized Prostate Cancer (Experimental): Patients with known localized prostate cancer with a soft tissue lesion at least 6mm or greater.
  Interventions: Drug: 18F DCFBC
- Biochemical Recurrence (Experimental): Patients with biochemical prostate cancer relapse after definitive treatment
  Interventions: Drug: 18F DCFBC
- Known Metastatic Disease (Experimental): Patients with identifiable metastatic disease on a conventional imaging modality. If only soft tissue metastasis, one lesion must measure 6mm or greater. Patients must have confirmation of prostate cancer prior to investigational imaging.
  Interventions: Drug: 18F DCFBC; Drug: Sodium (Na)18F positron emission tomography (PET)/computed tomography (CT)

INTERVENTIONS:
Drug: 18F DCFBC — Each subject will receive a single intravenous (i.v.) dose of 18F DCFBC by bolus injection at a rate of approximately 1 ml/3-5 sec.
Drug: Sodium (Na)18F positron emission tomography (PET)/computed tomography (CT)
  Other Names: Na 18F PET/CT
  Arms: Known Metastatic Disease

SUMMARY:
Background:

- Prostate cancer is the second leading cause of cancer deaths in American men. A chemical called a radiotracer helps doctors get images of this type of cancer. Researchers want to test a radiotracer called N-[N-[(S)-1,3-dicarboxypropyl]carbamoyl]-4-(18)F-fluorobenzyl-L-cysteine ((18)F-DCFBC) (18F-DCFBC).

Objective:

- To see if the radiotracer 18F-DCFBC can identify sites of prostate cancer in the body.

Eligibility:

- Men ages 18 and over with prostate cancer. The cancer must be newly diagnosed, have relapsed, or has spread outside the prostate.

Design:

* Participants will be screened with physical exam and medical history. They will give a blood sample.
* Participants will be divided into three groups.

Group 1: people with cancer only in the prostate scheduled for surgical prostate removal or biopsy at National Institutes of Health (NIH).

Group 2: people who had their prostate removed or had radiation therapy and now have a rising prostate-specific antigen (PSA) without other signs of disease.

Group 3: people whose cancer has spread to other areas of the body.

* Participants will have 18F-DCFBC injected into a vein then imaged in a positron emission tomography (PET)/computed tomography (CT) camera. During the scans, they will lie on their back on the scanner table.
* Group 1 will have a magnetic resonance imaging (MRI) scan. A tube will be placed in the rectum. Coils may be wrapped around the outside of the pelvis. Participants will have a contrast agent injected through an intravenous line.
* Group 3 will have another PET/CT scan with a different radiotracer, 18F NaF, within 21 days of the 18F-DCFBC scan to look for prostate cancer in the bone.
* Group 3 will repeat the two PET/CT scans 4-6 months after the initial scans.
* A few days after each scan, participants will be contacted for follow-up.

DETAILED DESCRIPTION:
Background

* Prostate cancer is the second leading cause of cancer deaths in American men.
* Current methods of imaging advanced prostate cancer (computed tomography ((CT) and bone scan) are non specific and new, more specific molecular imaging probes are sought.
* Many prostate cancers express the prostate specific membrane antigen (PSMA) a transmembrane protein with N-acetylated alpha-linked acidic dipeptidase (NAALADase) enzymatic activity. PSMA is also expressed in angiogenesis but otherwise has limited expression in normal tissue.
* N-[N-[(S)-1,3-dicarboxypropyl]carbamoyl]-4-(18)F-fluorobenzyl-L-cysteine ((18)F-DCFBC) (18F-DCFBC) is a radiolabeled positron emission tomography (PET) agent which binds with high affinity to PSMA and through whole-body non-invasive functional imaging, may provide new information on the expression of PSMA.

Primary Objective

- To assess the ability of 18F-DCFBC to differentiate between tumorous and nontumorous tissues in localized, recurrent (based on rising prostatic-specific antigen ((PSA) post treatment) and metastatic prostate cancer

Eligibility

* Subject is greater than or equal to 18 years old
* Eastern Cooperative Oncology Group (ECOG) 0-2 with adenocarcinoma of the prostate and fits criteria for one of the following:
* ARM 1

  -- Patients with known localized prostate cancer with a soft tissue lesion at least 6mm or greater.

  ---A multiparametric magnetic resonance imaging (MRI) (standard of care at the National Institutes of Health ((NIH) Clinical Center) must be performed within 4 months of18F-DCFBC injection with findings suggestive for prostate cancer and confirmed with histopathology.
* ARM 2

  * Patients with biochemical prostate cancer relapse after definitive treatment

    * For patients status post radiation therapy for prostate cancer, a PSA increase from post radiation therapy nadir
    * OR
    * For patients status post prostatectomy, any PSA >/=0.2 ng/ml
  * Nonspecific or no evidence for disease on standard imaging modality
* ARM 3

  * Patients with identifiable metastatic disease on a conventional imaging modality. If only soft tissue metastasis, one lesion must measure 6mm or greater. Patients must have confirmation of prostate cancer prior to 18F-DCFBC imaging.

Design

This is a single site 3-arm study enrolling a total of 110 evaluable patients: Arm 1 will include 12 patients with presumed localized prostate cancer scheduled to undergo prostatectomy or biopsy within 4 months of enrollment; Arm 2 will include 78 patients with biochemical recurrence without evidence of metastasis on conventional imaging; and Arm 3 will include 20 patients with known metastatic disease who may or may not be on or/scheduled to begin therapeutic intervention. Patients with presumed localized disease will undergo a standard of care, clinical multiparametric endorectal coil MRI in the National Cancer Institute (NCI) Molecular Imaging Clinic within 4 months of screening. Patients in Arm 3 will undergo 2 imaging sessions: baseline and 4-6 month follow-up. Clinical records (including PSA) and treatment (if any) that occurred in the imaging interval must be available. All patients in Arm 3 will also undergo Na18F PET/CT for evaluation of bone metastases as part of this protocol. In order to allow for a small number of nonevaluable patients, the accrual ceiling will be set at 125.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subject is greater than or equal to18 years old
* Platelet count > 50,000/mm^3
* Eastern Cooperative Oncology Group (ECOG) Performance score of 0 to 2.
* Ability to provide informed consent. All subjects must sign an informed consent form indicating their understanding of the investigational nature and risks of the study before any protocol-related studies are performed.
* Categories

  * ARM 1 only

    ---For patients with presumed localized disease (any tumor (T), nodes 0 (N0), metastasized 0 (M0)), a multiparametric magnetic resonance imaging (MRI) (standard of care at the National Institutes of Health ((NIH) Clinical Center) must be performed within 4 months of the N-[N-[(S)-1,3-dicarboxypropyl]carbamoyl]-4-(18)F-fluorobenzyl-L-cysteine ((18)F-DCFBC) (18F-DCFBC) injection with findings suggestive for prostate cancer and a prostate lesion at least 6mm or greater. Must have histopathologic confirmation of prostate cancer prior to 18F-DCFBC imaging.
  * ARM 2 only:

    * For patients status post radiation therapy for prostate cancer, any prostatic-specific antigen (PSA) increase from post radiation therapy nadir
    * OR
    * For patients status post prostatectomy, a PSA >/=0.2 ng/ml
    * Nonspecific or no evidence for disease on standard imaging modality
  * ARM 3 only:

    * Patients must have identifiable metastatic disease on at least 1 clinically indicated imaging modality. If only soft tissue metastasis, one lesion must measure at least 6mm or greater. Patients must have confirmation of prostate cancer prior to 18FDCFBC imaging

Note: A patient who is eligible for one arm, subsequently may cross-over into a different arm.

EXCLUSION CRITERIA:

* Subjects for whom participating would significantly delay the scheduled standard of care therapy
* Subjects with any coexisting medical or psychiatric condition that is likely to interfere with study procedures and/or results.
* Subjects with severe claustrophobia unresponsive to oral anxiolytics
* Other medical conditions deemed by the principal investigator (or associates) to make the subject unsafe/ineligible for protocol procedures.
* Subjects weighing > 350 lbs. (weight limit for scanner table), or unable to fit within the imaging gantry
* Serum creatinine > 2 times the upper limit of normal
* Total bilirubin > 2 times the upper limit of normal
* Liver transaminases (alanine aminotransferase (ALT), aspartate aminotransferase (AST)) greater than 3 times the upper limit of normal

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2014-07-12 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Liza Lindenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mena E, Lindenberg ML, Shih JH, Adler S, Harmon S, Bergvall E, Citrin D, Dahut W, Ton AT, McKinney Y, Weaver J, Eclarinal P, Forest A, Afari G, Bhattacharyya S, Mease RC, Merino MJ, Pinto P, Wood BJ, Jacobs P, Pomper MG, Choyke PL, Turkbey B. Clinical impact of PSMA-based 18F-DCFBC PET/CT imaging in patients with biochemically recurrent prostate cancer after primary local therapy. Eur J Nucl Med Mol Imaging. 2018 Jan;45(1):4-11. doi: 10.1007/s00259-017-3818-x. Epub 2017 Sep 11. PMID 28894899
- [Result] Turkbey B, Mena E, Lindenberg L, Adler S, Bednarova S, Berman R, Ton AT, McKinney Y, Eclarinal P, Hill C, Afari G, Bhattacharyya S, Mease RC, Merino MJ, Jacobs PM, Wood BJ, Pinto PA, Pomper MG, Choyke PL. 18F-DCFBC Prostate-Specific Membrane Antigen-Targeted PET/CT Imaging in Localized Prostate Cancer: Correlation With Multiparametric MRI and Histopathology. Clin Nucl Med. 2017 Oct;42(10):735-740. doi: 10.1097/RLU.0000000000001804. PMID 28806263
- [Result] Harmon SA, Bergvall E, Mena E, Shih JH, Adler S, McKinney Y, Mehralivand S, Citrin DE, Couvillon A, Madan RA, Gulley JL, Mease RC, Jacobs PM, Pomper MG, Turkbey B, Choyke PL, Lindenberg ML. A Prospective Comparison of 18F-Sodium Fluoride PET/CT and PSMA-Targeted 18F-DCFBC PET/CT in Metastatic Prostate Cancer. J Nucl Med. 2018 Nov;59(11):1665-1671. doi: 10.2967/jnumed.117.207373. Epub 2018 Mar 30. PMID 29602821
- [Derived] Rowe LS, Harmon S, Horn A, Shankavaram U, Roy S, Ning H, Lindenberg L, Mena E, Citrin DE, Choyke P, Turkbey B. Pattern of failure in prostate cancer previously treated with radical prostatectomy and post-operative radiotherapy: a secondary analysis of two prospective studies using novel molecular imaging techniques. Radiat Oncol. 2021 Feb 10;16(1):32. doi: 10.1186/s13014-020-01733-x. PMID 33568190
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0140.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Suspected Localized Prostate Cancer: Patients with known localized prostate cancer with a soft tissue lesion at least 6mm or greater.
  N-[N-[(S)-1,3-dicarboxypropyl]carbamoyl]-4-(18)F-fluorobenzyl-L-cysteine ((18)F-DCFBC) (18F DCFBC): Each subject will receive a single intravenous (i.v.) dose of 18F DCFBC by bolus injection at a rate of approximately 1 ml/3-5 sec.
Period: Overall Study
Arm/Group | Suspected Localized Prostate Cancer | Biochemical Recurrence | Known Metastatic Disease
Started | 16 | 69 | 31
Completed | 13 | 69 | 28
Not Completed | 3 | 0 | 3
Not completed — Withdrawal consent | 1 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Refused further treatment | 0 | 0 | 1
Not completed — Screening failure | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Suspected Localized Prostate Cancer | Biochemical Recurrence | Known Metastatic Disease | Total
Number analyzed (Participants) | 16 | 69 | 31 | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 34 | 14 | 54
  >=65 years | 10 | 35 | 17 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.58 (8.53) | 65.33 (6.67) | 63.93 (11.41) | 64.85 (8.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 16 | 69 | 31 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 69 | 31 | 116
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 7 | 3 | 14
  White | 12 | 59 | 27 | 98
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 69 | 31 | 116
Gleason Grade at Diagnosis [Count of Participants; unit: Participants] — Gleason grades help determine a good or bad prognosis for a with prostate cancer. Grade 5-6 are low on the scale and can indicate a less aggressive cancer. A higher number such as Grade 7-10 means a more aggressive cancer.
  Participants
    Gleason Grade 5 | 1 | 1 | 0 | 2
    Gleason Grade 6 | 3 | 7 | 7 | 17
    Gleason Grade 7-8 | 9 | 48 | 11 | 68
    Gleason Grade 9-10 | 3 | 12 | 9 | 24
    Not available | 0 | 1 | 1 | 2
Prior Prostate Cancer Therapy [Count of Participants; unit: Participants] — Androgen deprivation therapy (ADT). Radium 223 (Ra223).
  Participants
    None | 15 | 0 | 4 | 19
    Radical Prostatectomy | 0 | 49 | 1 | 50
    Brachytherapy/Radiation | 1 | 8 | 2 | 11
    ADT + Surgery or Radiation | 0 | 2 | 5 | 7
    ADT + Chemotherapy | 0 | 0 | 7 | 7
    ADT | 0 | 0 | 1 | 1
    Combo radical prostectomy and radiation therapy | 0 | 9 | 8 | 17
    Unknown | 0 | 1 | 0 | 1
Baseline Imaging [Count of Participants; unit: Participants] — N-[N-[(S)-1,3-dicarboxypropyl]carbamoyl]-4-(18)F-fluorobenzyl-L-cysteine ((18)F-DCFBC) Positron emission tomography (PET) Computed tomography (CT)
  Participants
    NaF PET/CT | 13 | 0 | 28 | 41
    DCFBC(1h) PET/CT | 13 | 68 | 28 | 109
    DCFBC(2h) PET/CT | 13 | 68 | 27 | 108
Prostatic-Specific Antigen (PSA) at Baseline [Median (Full Range); unit: ng/ml] — Normal PSA is defined as less than 4.0 ng/ml.
  ng/ml | 37.5 [3.26 to 216] | 1.63 [0.2 to 37.4] | 1.90 [0.01 to 4379] | 13.67 [1.15 to 1544]
Castration Status [Count of Participants; unit: Participants] — Castrate sensitive is defined as cancer that is outside the boundary of the prostate. Castrate resistant is defined as cancer of the prostate that no longer responds to one of the most common types of prostate treatment known as androgen deprivation therapy (ADT) (i.e. lowers testosterone levels).
  Participants
    Untreated | 0 | 0 | 3 | 3
    Castrate-sensitive | 0 | 0 | 14 | 14
    Castrate-resistant | 0 | 0 | 11 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Local Recurrence, Lymph Node Metastases or Distant Metastatic Sites Detected by N-[N-[(S)-1,3-dicarboxypropyl]Carbamoyl]-4-(18)F-fluorobenzyl-L-cysteine ((18)F-DCFBC) Imaging
Description: Any abnormal focus of 18F-DCFBC uptake higher than the surrounding background and not associated with physiological uptake was considered positive for prostate cancer, and each was classified as local recurrence, lymph node metastases or distant metastatic sites.
Time Frame: 1 hour and 2 hour timepoints at baseline
Population: In Arm 1: 3 patients were excluded from analysis due to prior focal ablation therapy (1), prior brachytherapy (1), and lack of histopathologic confirmation tissue.
  Arm 2: 1 patient had technical issues and was not included in the final analysis Arm 3: 2 patients were not imaged and 1 patient withdrew consent
Measure: Count of Participants; unit: Participants
Arm/Group | Suspected Localized Prostate Cancer | Biochemical Recurrence | Known Metastatic Disease
Number analyzed (Participants) | 13 | 68 | 28
Participants
  Lymph nodes | 1 | 39 | 28
  Distant sites | 0 | 10 | 10
  Prostate bed/anastomosis | 8 | 30 | 28

2. Primary Outcome: Number of Lesions Detected by N-[N-[(S)-1,3-dicarboxypropyl]Carbamoyl]-4-(18)F-fluorobenzyl-L-cysteine ((18)F-DCFBC)
Description: Any abnormal focus of 18F-DCFBC uptake higher than the surrounding background and not associated with physiological uptake was considered a positive lesion for prostate cancer.The measure would be compared with other imaging or pathology.
Time Frame: 1 hour and 2 hour timepoints at baseline
Population: as for outcome 1
Measure: Number; unit: lesions
Arm/Group | Suspected Localized Prostate Cancer | Biochemical Recurrence | Known Metastatic Disease
Number analyzed (Participants) | 13 | 68 | 28
lesions | 9 | 79 | 140

3. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 42 months and 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | Suspected Localized Prostate Cancer | Biochemical Recurrence | Known Metastatic Disease
Number analyzed (Participants) | 16 | 69 | 31
Participants | 1 | 3 | 8

4. Secondary Outcome: Number of Detectable Lesions in Bone With Respect to 18F-DCFBC Imaging and/or Na18F Positron Emission Tomography (PET)/Computed Tomography (CT) in Patients With Known Metastatic Disease
Description: 18F-DFBC and conventional imaging was used to identify positive lesions in bone.
Time Frame: 3 months
Population: The Suspected Localized Prostate Cancer and Biochemical Recurrence Arms/Groups are not applicable for this outcome measure, thus are not represented here. Data was collected for 31 participants but only 28 had data evaluable for final analysis in the Known Metastatic Group.
Measure: Number; unit: number of bone lesions
Units Other Than Participants: lesions
Arm/Group | Known Metastatic Disease
Number analyzed (Participants) | 28
Number analyzed (lesions) | 241
number of bone lesions | 185

5. Secondary Outcome: Average Standardized Uptake Value (SUVmax) for Primary Prostate Cancer Patients Compared to Benign Prostatic Hyperplasia (BPH)
Description: Primary prostate cancer was compared to BPH nodules and normal prostate tissue using a one-way analysis of variance (Anova). Negative uptake is defined as tumor uptake less than adjacent background soft tissue, or blood pool for lymph nodes.
Time Frame: 1 hour and 2 hour post injection (p.i.)
Population: 3 patients were excluded from analysis due to prior focal ablation therapy (1), prior brachytherapy (1), and lack of histopathologic confirmation tissue. The Biochemical Recurrence and Known Metastatic Disease Arms/Groups are not applicable for this outcome measure, thus are not represented here.
Measure: Mean (Standard Deviation); unit: standardized uptake value (SUV)
Arm/Group | Suspected Localized Prostate Cancer
Number analyzed (Participants) | 13
standardized uptake value (SUV)
  Primary prostate tumor - 1 hour post injection | 5.8 (4.4)
  BPH nodules - 1 hour post injection | 2.1 (0.3)
  Normal prostate - 1 hour post injection | 2.1 (0.4)
  Primary prostate tumor - 2 hour post injection | 5.9 (5.3)
  BPH nodules - 2 hour post injection | 2.0 (0.36)
  Normal prostate tumor - 2 hour post injection | 2.0 (0.28)
Statistical Analysis 1: Comparison: Suspected Localized Prostate Cancer; At 1 hour post injection; Test type: Other; p = 0.0033, ANOVA
Statistical Analysis 2: Comparison: Suspected Localized Prostate Cancer; At 2 hour post injection; Test type: Other; p = 0.012, ANOVA

6. Secondary Outcome: Median Tumor Foci Size in Suspected Localized Prostate Cancer Patients Undergoing Prostatectomy
Description: Tissue was obtained and stained with hematoxylin-eosin. The resulting whole mount specimens were correlated with MRI and PET/CT imaging. For each dominant/index tumor (largest tumor with highest Gleason score) was determined.
Time Frame: 1 month
Population: 3 patients were excluded from analysis, because of prior focal laser ablation therapy (n=1), prior brachytherapy (n=1), and lack of histopathology confirmation tissue (n=1). The Biochemical Recurrence and Known Metastatic Disease Arms/Groups are not applicable for this outcome measure, thus are not represented here.
Measure: Median (Full Range); unit: cm
Units Other Than Participants: Tumor foci
Arm/Group | Suspected Localized Prostate Cancer
Number analyzed (Participants) | 13
Number analyzed (Tumor foci) | 25
cm | 1.5 [0.6 to 4.7]
Statistical Analysis 1: Comparison: Suspected Localized Prostate Cancer; Test type: Equivalence — One way analysis variance; p < 0.05, variance

7. Secondary Outcome: Detectability of Suspicious Prostate Cancer Lesions in Suspected Localized Prostate Cancer Patients With Prostate Gland
Description: Visualizing positive lesions with DCFBC and mpMRI.
Time Frame: 3 months
Population: as for outcome 6
Measure: Number; unit: percent of lesions identified
Units Other Than Participants: lesions
Arm/Group | Suspected Localized Prostate Cancer
Number analyzed (Participants) | 13
Number analyzed (lesions) | 25
percent of lesions identified
  18F-DCFBC | 36
  mpMRI | 96

8. Secondary Outcome: Detectability of Suspicious Tumors Based on Prostate Specific-Antigen (PSA) Levels in the Biochemical Recurrence Group
Description: Visualizing positive lesions as a function of PSA value. Undetectable PSA is normal in this population.
Time Frame: 3 months
Population: 1 patient had technical issues and was not included in the final analysis.
Measure: Number; unit: percent of tumors identified
Arm/Group | Biochemical Recurrence
Number analyzed (Participants) | 68
percent of tumors identified
  <0.5 ng/mL | 15
  0.5 to <1.0 ng/mL | 46
  1.0 to 2.0 ng/mL | 83
  2.0 ng/mL | 77

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 42 months and 21 days.
Groups:
- Suspected Localized Prostate Cancer: Patients with known localized prostate cancer with a soft tissue lesion at least 6mm or greater.
  N-[N-[(S)-1,3-dicarboxypropyl]carbamoyl]-4-(18)F-fluorobenzyl-L-cysteine ((18)F-DCFBC) (18F DCFBC: Each subject will receive a single intravenous (i.v.) dose of 18F DCFBC by bolus injection at a rate of approximately 1 ml/3-5 sec.
Arm/Group | Suspected Localized Prostate Cancer | Biochemical Recurrence | Known Metastatic Disease
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/69 | 2/31
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/69 | 4/31
Other Adverse Events (participants affected / at risk) | 1/16 | 3/69 | 8/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suspected Localized Prostate Cancer (N=16) | Biochemical Recurrence (N=69) | Known Metastatic Disease (N=31)
Gastrointestinal disorders - Other, nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Death NOS (General disorders) | 0 (0) | 0 (0) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Death due to progressive disease
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suspected Localized Prostate Cancer (N=16) | Biochemical Recurrence (N=69) | Known Metastatic Disease (N=31)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other, near syncope (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-12-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT02190279/Prot_SAP_000.pdf
  • Informed Consent Form (2015-12-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT02190279/ICF_001.pdf